CLINICAL TRIAL: NCT04625595
Title: A Phase 1b, Randomized, Single-blind, Placebo-controlled, Multiple Ascending Dose (MAD) Study to Assess the Steady-State Pharmacokinetics and DQ8 Blocking Efficacy of Orally Administered IMT-002 in Patients With Type 1 Diabetes and HLA-DQ8
Brief Title: Multiple Ascending Dose (MAD) Study of IMT-002 in HLA-DQ8-positive Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunomolecular Therapeutics, Inc. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT-002-0102
Record Dates: First submitted 2020-10-20; First posted 2020-11-12 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-06

CONDITIONS: Type1 Diabetes
Keywords: diabetes; prescreening; autoimmunity; HLA
MeSH Terms: conditions — Diabetes Mellitus; Autoimmune Diseases | interventions — BID protein, human; Capsules; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 350 mg BID (700 mg total daily dose) of active drug or placebo (Experimental): Low dose, drug IMT-002
  Interventions: Drug: 350mg BID (700mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule
- 1050 mg QD (1050 mg total daily dose) of active drug or placebo (Experimental): Moderate dose, drug IMT-002
  Interventions: Drug: 1050mg QD (1050mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule
- 700 mg BID (1400 mg total daily dose) of active drug or placebo (Experimental): Moderate to high dose, drug IMT-002
  Interventions: Drug: 700mg BID (1400mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule
- 1050 mg BID (2100 mg total daily dose) of active drug or placebo (Experimental): High dose, drug IMT-002
  Interventions: Drug: 1050mg BID (2100mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule

INTERVENTIONS:
Drug: 350mg BID (700mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule — Oral drug or placebo self-administered by subject as a capsule by mouth once-daily or twice-daily
  Other Names: 350mg BID
  Arms: 350 mg BID (700 mg total daily dose) of active drug or placebo
Drug: 700mg BID (1400mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule — Oral drug or placebo self-administered by subject as a capsule by mouth once-daily or twice-daily
  Other Names: 700mg BID
  Arms: 700 mg BID (1400 mg total daily dose) of active drug or placebo
Drug: 1050mg QD (1050mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule — Oral drug or placebo self-administered by subject as a capsule by mouth once-daily or twice-daily
  Other Names: 1050mg QD
  Arms: 1050 mg QD (1050 mg total daily dose) of active drug or placebo
Drug: 1050mg BID (2100mg total daily) IMT-002, D-methyldopa, active formulation in capsule or Placebo, microcrystalline cellulose in capsule — Oral drug or placebo self-administered by subject as a capsule by mouth once-daily or twice-daily
  Other Names: 1050mg BID
  Arms: 1050 mg BID (2100 mg total daily dose) of active drug or placebo

SUMMARY:
This study is designed to characterize the safety, steady-state pharmacokinetics (PK) of IMT-002, and will serve as a dose range identification for the pharmacodynamic effect of blocking self-antigen presentation in adults with type 1 diabetes (T1D) having the human leukocyte antigen (HLA)-DQ8 gene.

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo-controlled study that will include 4 ascending dose cohorts: 350 mg twice daily (BID), 1050 mg once daily (QD), 700 mg BID, and 1050 mg BID. Subjects will undergo prescreening for genetic typing and then screening procedures up to 28 days prior to the first dose to determine eligibility. T1D adults between 18 and 45 years of age, inclusive, who are positive for at least one gene encoding for HLA-DQ8 (DQA1*0301, DQB1*0302) will be enrolled.

Each cohort will include 6 subjects on active drug, and the study will include 6 subjects total on placebo. Each cohort will participate in a 2-week dosing period. Enrollment of the cohorts will be sequentially staggered such that initial safety data after the first four subjects assigned to active treatment complete one week of treatment in each cohort will be reviewed before the next ascending dose cohort is enrolled. The safety reviews will include cumulative safety data for all subjects to that point. Subjects will have 5 scheduled clinic visits: screening, first day of dosing, 1 week after dosing begins, 2 weeks after dosing begins (end of treatment), and 1 week following the final dose. Subjects will self-administer study drug on non-clinic treatment days. Safety assessments will be conducted at all study visits. Insulin use (dose and frequency) will be monitored.

Pharmacokinetic (PK) assessments will be evaluated at every visit during the treatment period to characterize the following: single dose PK, trough PK and steady PK. Pharmacodynamic (PD) and immunological assessments will be evaluated before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the ICF as described in Appendix 3 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Man or woman, 18 to 45 years of age inclusive at the time of signing the ICF.
3. Has received a diagnosis of T1D according to the criteria from the American Diabetes Association.
4. Positive for at least one gene encoding for HLA-DQ8 (DQB*0302).
5. If male, and of reproductive potential, willing to use medically acceptable birth control (Appendix 5), unless the female partner is postmenopausal or surgically sterile, until study completion and for at least 30 days after the last dose of study treatment and refrain from donating sperm during this period.
6. If female: (a) surgically sterile or (b) postmenopausal or (c) if of reproductive potential, willing to use medically acceptable birth control (eg, female hormonal contraception, barrier methods or sterilization (Appendix 5) until study completion and for at least 30 days (one menstrual cycle).

Exclusion Criteria:

1. Inability or unwillingness of a subject to give written informed consent or comply with the study protocol.
2. No HLA-DQ8 gene (DQB*03:02).
3. Any of the following hematologic abnormalities at the time of screening, confirmed by repeat tests:

   1. Leukopenia (<3,000 leukocytes/μL)
   2. Neutropenia (<1,500 neutrophils/μL)
   3. Thrombocytopenia (<125,000 platelets/μL)
   4. Hemoglobin less than 10 g/dl
4. Evidence of liver dysfunction, with ALT > 2.5 times the upper limit of normal (ULN) or AST >3.0 times ULN persistent for 1 week or greater.
5. Evidence of renal insufficiency as indicated by serum creatinine of >1.5 times ULN, confirmed by a repeat test.
6. Clinically significant abnormal physical examination, vital signs, or 12-lead ECG at screening as deemed appropriate by the investigator.
7. Has a history of or current clinically significant medical illness including, but not limited to, cardiac arrhythmias or other cardiac disease; significant pulmonary disease; neurologic or psychiatric disease; infection; or any other illness that the investigator considers should exclude the subject or that could interfere with the interpretation of the study results.
8. Body mass index (BMI) > 32 kg/m2.
9. Unstable blood sugar control defined as one or more episodes of severe hypoglycemia (defined as hypoglycemia that required the assistance of another person) within the last 30 days.
10. Use of a treatment that is known to cause a significant, ongoing change in the course of T1D or immunologic status, within 4 weeks prior to participation; this includes high-dose inhaled, extensive topical or systemic glucocorticoids.
11. History of any organ transplant, including islet cell transplant.
12. Pregnant or anticipates pregnancy during the 2-week study period or within 30 days following the last dose of study drug.
13. Use of investigational drugs within 90 days of participation.
14. Currently taking methyldopa (Aldomet) at the time of randomization or taken within the past 3 months.
15. Currently taking ferrous sulfate or ferrous gluconate, which are indicated for the treatment of anemia (hematological disease), or taken within the past 30 days.
16. Unable to avoid medications that affect stomach pH, such as proton pump inhibitors or histamine H2 receptor blockers.
17. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the Investigator, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.
18. Has a history of the human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or another clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
19. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.
20. Has preplanned surgery or procedures that would interfere with the conduct of the study.
21. Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Treatment and follow-up period, Day 21
  Frequency tabulated as number of participants with adverse and serious adverse events (AEs)
Change from baseline in electrocardiogram (ECG) | Day 1, Day 7, Day 14 and Day 21
  Single 12-lead ECG will be measured in a supine position after 5 minutes rest and measure QRS, QT, and QTc intervals
Change in total daily insulin use | Day 1, Day 7, Day 14 and Day 21
  At each study visit, total daily insulin (ie, total insulin administered over the previous 24-hour period) will be entered in the Concomitant Medications CRF

SECONDARY OUTCOMES:
Pharmacokinetic (PK) measurement in blood plasma, Cmax | Day 1, Day 7, Day 14
  Cmax, maximum plasma concentration during a dosing interval
Cytokine level from in vitro presentation of antigen by HLA-DQ8 | Day 1, Day 7, Day 14 and Day 21
  Change from baseline of cytokine, interleukin-2, level produced in T-cell based in vitro assay of blood sample resulting from presentation of insulin or gluten peptide antigen by HLA-DQ8

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Prosciento, Inc., Chula Vista, California
  - Barbara Davis Center, Aurora, Colorado
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrov DA, Alkanani A, McDaniel KA, Case S, Baschal EE, Pyle L, Ellis S, Pollinger B, Seidl KJ, Shah VN, Garg SK, Atkinson MA, Gottlieb PA, Michels AW. Methyldopa blocks MHC class II binding to disease-specific antigens in autoimmune diabetes. J Clin Invest. 2018 May 1;128(5):1888-1902. doi: 10.1172/JCI97739. Epub 2018 Apr 3. PMID 29438107
- [Background] Ostrov DA, Gottlieb PA, Michels AW. Rationally designed small molecules to prevent type 1 diabetes. Curr Opin Endocrinol Diabetes Obes. 2019 Apr;26(2):90-95. doi: 10.1097/MED.0000000000000470. PMID 30694829
- [Background] Au WY, Dring LG, Grahame-Smith DG, Isaac P, Williams RT. The metabolism of 14 C-labelled -methyldopa in normal and hypertensive human subjects. Biochem J. 1972 Aug;129(1):1-10. doi: 10.1042/bj1290001. PMID 4646774
- [Background] GILLESPIE L Jr, OATES JA, CROUT JR, SJOERDSMA A. Clinical and chemical studies with alpha-methyl-dopa in patients with hypertension. Circulation. 1962 Feb;25:281-91. doi: 10.1161/01.cir.25.2.281. No abstract available. PMID 13898638
- [Background] SJOERDSMA A, VENDSALU A, ENGELMAN K. STUDIES ON THE METABOLISM AND MECHANISM OF ACTION OF METHYLDOPA. Circulation. 1963 Oct;28:492-502. doi: 10.1161/01.cir.28.4.492. No abstract available. PMID 14068757